CLINICAL TRIAL: NCT05197166
Title: Baropodometric Assessment of the Podiatric Profile of Nursing Students in Clinical Settings
Status: Completed | Type: Observational
Sponsor: Escola Superior de Enfermagem de Coimbra (Other)
Collaborators: University of Turku (Other); Universidade Católica Portuguesa (Other)
Responsible Party: Principal Investigator, Rafael Alves Bernardes, Registered Nurse, Escola Superior de Enfermagem de Coimbra
Other Study IDs: 151102
Record Dates: First submitted 2021-12-15; First posted 2022-01-19 (Actual); Last update posted 2023-09-14 (Actual); Status verified 2023-09

CONDITIONS: Foot Diseases; Ankle Disorders Injuries
Keywords: foot disorders; ankle disorders; nursing; foot health; foot self-care
MeSH Terms: conditions — Foot Diseases; Ankle Injuries

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Nursing students: Nursing students exposed to standing environments (prolonged walking and prolonged standing) during acute clinical settings (e.g., hospitals).
  Interventions: Other: Acute Clinical Settings

INTERVENTIONS:
Other: Acute Clinical Settings — Acute clinical settings, like hospitals, where students are exposed to normal daily shift activities, involving prolonged walking and standing positions.

SUMMARY:
The nursing profession is highly affected by exhausting positions, namely prolonged standing and walking, which are the second work-related factor hindering foot health. In fact, the most common work-related disorders among nurses and nursing students are those related to lower limbs, particularly the foot and ankle. Such disorders, if not adequately prevented, contribute to the decrease in quality of life and high student drop-out rates.

To effectively develop preventive interventions among students, namely self-care actions, it's important to assess with detail the relationship and influence that clinical settings have on foot health. According to some authors, the biomechanics of many foot disorders are still poorly understood, and more studies are needed.

In this sense, the aim of this study is to understand the influence of prolonged standing and walking positions on nursing students' foot health. Moreover, what's the relationship between the podiatric profile (regional force and pressure exerted on the foot) and related signs and symptoms.

DETAILED DESCRIPTION:
Work-related injuries, particularly musculoskeletal injuries, are usually an important cause of decreased quality of life and absenteeism from work, being very common in the nursing profession and also among students. Among the most common injuries are those related to the lower limbs, particularly feet and ankles, and the foot health of nurses is not satisfactory, with a great shortage of specific studies in this area and in this population.

Although several studies identify this problem, few describe in detail the causes of pain or discomfort. On the other hand, the podiatry evaluations are poor, which limits a more detailed knowledge of the phenomenon under study. Some solutions, namely the development of ergonomic footwear are insufficient and few interventions are adequate to improve the foot health of nursing students.

The present study aims to understand the influence of prolonged standing and walking positions on nursing students' foot health. Moreover, what's the relationship between the podiatric profile (regional force and pressure exerted on the foot) and related signs and symptoms.

The observational study will consist of two moments (before and after clinical setting periods), in which the participants (Nursing students) will complete a four-dimensional foot health self-assessment instrument (skin health, nail health, foot structure, pain). Additionally, the podiatric profile will be assessed through a force platform scan, which will score force and pressure values. Moreover, foot posture and foot function will be evaluated, through the modified arch index (MAI) and pressure excursion index (CPEI), respectively. Relevant variables will include spatio-temporal, kinematic, and kinetic data.

ELIGIBILITY:
Inclusion Criteria:

* A nursing student enrolled in a learning acute clinical setting (e.g., hospitals).
* No diagnosed chronic systematic diseases (e.g., rheumatoid arthritis).
* No diagnosed metabolic disorders (e.g., diabetes).
* No visible lower limb swelling.
* No venous or lymphatic insufficiency.
* Voluntary written consent.

Exclusion Criteria:

* Presence of contraindications for baropodometric-related measurements;
* No consent to take part in the study.
* History of orthopaedic, neurological, and/or musculoskeletal problems likely to affect gait.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Nursing students (enrolled in a nursing bachelor of a Nursing School), in learning clinical settings (acute care),
Sampling Method: Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2022-01-01 (Actual); Primary Completion 2022-07-26 (Actual); Study Completion 2022-12-30 (Actual)

PRIMARY OUTCOMES:
Change in Podiatric Profile at 5 months | Evaluated before (Month 0) and after (Month 5) the exposure (acute clinical settings).
  It relates to specific foot-related dynamic variables while standing or walking, illustrating the actual behaviour of the foot during activity. The podiatric profile is assessed through a pedography platform, which gives values of pressure (throughout time), exerted force, and contact areas of the foot.
Change in Foot Health at 5 months | Evaluated before (Month 0) and after (Month 5) the exposure (acute clinical settings).
  Foot health relates to the observed clinical parameters, signs, and symptoms of this body part, namely skin, nails, and structure, and is evaluated through a subjective self-assessment Liker-type instrument with four dimensions related to general foot health.

SECONDARY OUTCOMES:
Foot Self-Care Knowledge | During the exposure time; between Month 0 and Month 5.
  Self-care knowledge is assessed through a four-dimensional questionnaire, where specific interventions for the promotion and prevention of foot and ankle disorders are evaluated.
Student's perceptions | After exposure time (Month 5).
  Nursing student's perceptions on the influence of foot health in their quality of life during exposure time. It is evaluated through semi-structured interviews and focus groups.

CONTACTS AND LOCATIONS:
Locations (1):
- Nursing School of Coimbra (ESEnfC), Coimbra, Portugal

IPD SHARING:
Plan to Share IPD: No
IPD will not be shared with other researchers

REFERENCES:
- [Background] Stolt M, Miikkola M, Suhonen R, Leino-Kilpi H. Nurses' Perceptions of Their Foot Health: Implications for Occupational Health Care. Workplace Health Saf. 2018 Mar;66(3):136-143. doi: 10.1177/2165079917727011. Epub 2017 Aug 31. PMID 28856977
- [Background] Stolt M, Katajisto J, Peltonen J, Suhonen R, Leino-Kilpi H. Development and testing of a new electronic foot health promotion programme on nurses' foot self-care. BMC Nurs. 2020 Apr 19;19:29. doi: 10.1186/s12912-020-00423-z. eCollection 2020. PMID 32327936
- [Background] Bakker EJM, Verhaegh KJ, Kox JHAM, van der Beek AJ, Boot CRL, Roelofs PDDM, Francke AL. Late dropout from nursing education: An interview study of nursing students' experiences and reasons. Nurse Educ Pract. 2019 Aug;39:17-25. doi: 10.1016/j.nepr.2019.07.005. Epub 2019 Jul 15. PMID 31352089
- [Background] Hagedorn TJ, Dufour AB, Riskowski JL, Hillstrom HJ, Menz HB, Casey VA, Hannan MT. Foot disorders, foot posture, and foot function: the Framingham foot study. PLoS One. 2013 Sep 5;8(9):e74364. doi: 10.1371/journal.pone.0074364. eCollection 2013. PMID 24040231
- [Background] Chiwaridzo M, Makotore V, Dambi JM, Munambah N, Mhlanga M. Work-related musculoskeletal disorders among registered general nurses: a case of a large central hospital in Harare, Zimbabwe. BMC Res Notes. 2018 May 18;11(1):315. doi: 10.1186/s13104-018-3412-8. PMID 29776452
- [Background] Stolt M, Suhonen R, Puukka P, Viitanen M, Voutilainen P, Leino-Kilpi H. Nurses' knowledge of foot care in the context of home care: a cross-sectional correlational survey study. J Clin Nurs. 2015 Oct;24(19-20):2916-25. doi: 10.1111/jocn.12922. Epub 2015 Jul 14. PMID 26179162
- [Background] Stolt M, Suhonen R, Kielo E, Katajisto J, Leino-Kilpi H. Foot health of nurses-A cross-sectional study. Int J Nurs Pract. 2017 Aug;23(4). doi: 10.1111/ijn.12560. Epub 2017 Jun 19. PMID 28631438
- [Background] Yan P, Li F, Zhang L, Yang Y, Huang A, Wang Y, Yao H. Prevalence of Work-Related Musculoskeletal Disorders in the Nurses Working in Hospitals of Xinjiang Uygur Autonomous Region. Pain Res Manag. 2017;2017:5757108. doi: 10.1155/2017/5757108. Epub 2017 Jul 13. PMID 28785160
- [Background] Richardson A, Gurung G, Derrett S, Harcombe H. Perspectives on preventing musculoskeletal injuries in nurses: A qualitative study. Nurs Open. 2019 Apr 13;6(3):915-929. doi: 10.1002/nop2.272. eCollection 2019 Jul. PMID 31367415
- [Background] Sanchez-Saez JM, Palomo-Lopez P, Becerro-de-Bengoa-Vallejo R, Calvo-Lobo C, Losa-Iglesias ME, Lopez-Del-Amo-Lorente A, Lopez-Lopez D. Stability of Three Different Sanitary Shoes on Healthcare Workers: A Cross-Sectional Study. Int J Environ Res Public Health. 2019 Jun 16;16(12):2126. doi: 10.3390/ijerph16122126. PMID 31208123
- [Background] Abledu JK, Offei EB. Musculoskeletal disorders among first-year Ghanaian students in a nursing college. Afr Health Sci. 2015 Jun;15(2):444-9. doi: 10.4314/ahs.v15i2.18. PMID 26124790
- [Derived] Bernardes RA, Caldeira S, Parreira P, Sousa LB, Almeida IF, Santos-Costa P, Paiva-Santos F, Guardado Cruz A. Baropodometric Assessment of the Podiatric Profile of Nursing Students in Clinical Settings: A Study Protocol. Front Public Health. 2022 May 12;10:862048. doi: 10.3389/fpubh.2022.862048. eCollection 2022. PMID 35646767